CLINICAL TRIAL: NCT00935519
Title: Cementless New Alumina-zirconia(4th Generation Ceramic Bearing) Composite Ceramic Bearing Total Hip Arthroplasty (THA) in Asian Patients : a 10 Year Minimum Follow-up Study
Brief Title: Cementless New Alumina-zirconia Ceramic Bearing Total Hip Arthroplasty (THA) in Asian Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Kyung-Hoi Koo, Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNU 09-01
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: total hip arthroplasty, ceramic, survival

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ceramic bearing (Other): Survival rate of THA with use of the new alumina-zirconia(4th generation ceramic bearing) composite ceramic bearing at a minimum of 10 years follow-up.
  Interventions: Device: 4th generation ceramic bearing composite ceramic bearing

INTERVENTIONS:
Device: 4th generation ceramic bearing composite ceramic bearing — THA with use of the new alumina-zirconia(4th generation ceramic bearing) composite ceramic bearing at a minimum of 10 years follow-up.
  Other Names: delta ceramic

SUMMARY:
This study will evaluate a midterm clinical and radiologic outcome patients who undergo new alumina-zirconia composite ceramic bearing THA.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) using a metal-on-polyethylene articulation has become one of the most effective procedures for the surgical treatment for end-stage hip disease.

However, polyethylene wear debris-induced osteolysis has been postulated to cause/contribute to the aseptic loosening of a THA, and hence, is regarded to be an important factor in its in vivo longevity.

In the third generation of ceramic manufacturing, many improvements, such as hot isostatic pressing, laser marking, and non destructive proof-testing for all ceramic components, have been introduced. This third generation ceramic component has high purity, high density, and small grain size, and, therefore, has a very high potential for resisting crack propagation, which may culminate in its fracture. In spite of this, a number of substantial concerns, such as ceramic fracture, impingement-associated fatigue failure, wear, and osteolysis after long-term follow-up, persist with the use of ceramics in THA.

In addition, the third generation ceramic articulation is associated with an increased incidence of dislocation because ceramic liners with elevated rim and extended-long-neck ceramic heads are not available.

However, new alumina-zirconia composites bearing implants (4th generation ceramic bearing) affords various options such as large head and thin liner, which may decrease the ceramic fracture rate and dislocation rate and improve the longevity of THA. In addition, large head can improve the range of motion and possible traditional cross-legged sitting position of Koreans without impingement between the neck and liner rim.

So far, the patients who are underwent THA using 28 mm femoral head diameter complains limitation of range of motion and feeling impingement sensation at sitting on the floor with their legs crossed. There have been increasing complaints especially from Korean patients regarding the difficulties associated with carrying out their daily activities, whose life style involves sitting on the floor with their legs crossed. Therefore, large head of new alumina-zirconia composites bearing implants(4th generation ceramic bearing) expects increasing satisfaction of Korean patients.

This is the first study, to our knowledge, of an evaluation of clinical outcome of THA with use of the new alumina-zirconia(4th generation ceramic bearing) composite ceramic bearing and the functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have femoral head osteonecrosis
* Subjects who have primary or secondary osteoarthritis
* Subjects who have femoral neck fracture
* Subjects who have infection sequels
* Subjects who have rheumatoid arthritis or ankylosing spondylitis
* Subjects who have developmental dysplasia of the hip or acetabular dysplasia

Exclusion Criteria:

* Subjects who have active infection
* Subjects who have unstable medical illness
* Subjects who have rapidly progressive neurological disease
* Subjects who have revision surgery or bipolar endoprosthesis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2009-05; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Survival rate of THA with use of the new alumina-zirconia(4th generation ceramic bearing) composite ceramic bearing at a minimum of 10 years follow-up. | up to 10 years

SECONDARY OUTCOMES:
The performance in patients younger than 50 years at 10 years follow up | Follow-up evaluations will be performed at six weeks; at three, six, nine, and twelve months and every 12 months thereafter.
Evaluation between preoperative and postoperative of Harris hip score, UCLA activity score, WOMAC, and Subject satisfaction score at a minimum of 5 years follow-up. | Follow-up evaluations will be performed at six weeks; at three, six, nine, and twelve months and every 12 months thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Hoi Koo, professor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul national University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea